CLINICAL TRIAL: NCT06621004
Title: Low Dose Magnesium Sulphate in Nasal Surgery
Brief Title: Low Dose Magnesium Sulphate
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Assistant professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMASU R205/2024
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Mean Arterial Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- propranolol (Active Comparator): 1 mg propranolol will be prepared in a 10 ml syringe (100 ug/ml). Propranolol will be given 200-300 ug bolus followed by increments of 100 ug until MABP becomes 50-60 mmHg and HR 50 - 70 b/ m.
  Interventions: Drug: Patients will receive propranolol 1-2 mg.
- propranolol and magnesium sulphate (Active Comparator): 1g MgSo3 ampoule (10ml) will be prepared in a syringe pump to be given at a rate of 40 ml/hr in the group and 1 mg propranolol will be prepared in a 10 ml syringe (100 ug/ml). Propranolol will be given 200-300 ug bolus followed by increments of 100 ug until MABP becomes 50-60 mmHg and HR 50 - 70 b/ m.
  Interventions: Drug: Patients will receive propranolol 1-2 mg.; Drug: Patient receives magnesium sulphate

INTERVENTIONS:
Drug: Patients will receive propranolol 1-2 mg. — Patients will receive propranolol 1-2 mg. prepared in a 10 ml syringe (100 ug/ml).
Drug: Patient receives magnesium sulphate — Magnesium sulphate 10%: 1g ampoule (10ml), will be prepared in a syringe pump to be given at a rate of 40 ml/hr . Another syringe of 10 ml 0.9% sodium chloride will be prepared to be given in group (P).
  Arms: propranolol and magnesium sulphate

SUMMARY:
This clinical trial aims to compare Patients who receive propranolol 1-2 mg to Patients who receive propranolol 1-2 mg in addition to magnesium sulphate infusion 10 mg/kg to see if IV magnesium can stability mean arterial blood pressure and heart rate in patients undergoing nasal surgeries as well as the quality of postoperative analgesia, degree of sedation mean arterial blood pressure and HR will be recorded intraoperative and Participants will be asked to rate the pain at the first, second, fourth, sixth and 24th postoperative hour using the VAS score.

* Analgesic requirements: The time to first demand analgesia and the total amount of analgesia required in the 1st 24 will be recorded.
* Sedation score: the degree of sedation will be assessed using the Ramsy sedation score

DETAILED DESCRIPTION:
This prospective, randomized controlled clinical trial aims to establish the effect of magnesium sulphate during nasal surgery regarding deliberate hypotension, postoperative analgesia and sedation with minimal side effects.

this study will be conducted in the plastic surgery and ENT operating rooms at ASUH 130 patients undergoing rhinoplasty or functional endoscopic sinus surgery (FESS) operation under general anaesthesia.

patients will be allocated into 2 groups 65 patients each using a computer-generated randomization list.

Group (P): Patients will receive propranolol 1-2 mg. Group (PM): Patients will receive propranolol 1-2 mg in addition to magnesium sulphate infusion 10 mg/kg.

* ABP and HR are continuously monitored and will be recorded before the start of anaesthesia (T1), after intubation (T2), at skin incision (T3), at manipulation of nasal bones (T4), at extubation (T5), before discharge to PACU (T6), and after 30 min in PACU.
* Surgical duration (time from skin incision till skin closure).
* Extubation time (from the end of anaesthesia to extubation)
* Modified Alderete score will be assessed and recorded every 5 minutes until discharge. Patients will be discharged upon achieving an Aldrete score of ≥ 9.
* The time to discharge will be recorded.
* VAS score for pain:
* Analgesic requirements: The time to first demand analgesia and the total amount of analgesia required in the 1st 24 will be recorded.
* Sedation score: the degree of sedation will be assessed using the Ramsy sedation score where all be recorded

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing rhinoplasty or functional endoscopic sinus surgery (FESS) operation under general anesthesia
* ASA I or II
* Duration of surgery will be 1-2 hours

Exclusion Criteria:

* Hypertension,
* Myasthenia gravis or other muscular disease,
* Impaired kidney or liver functions,
* History of drug or alcohol abuse,
* History of antidepressant and calcium channel blocker use,
* Mental retardation and hysterical patients.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
mean arterial blood pressure | intraoperative
  mmHg

SECONDARY OUTCOMES:
analgesia | 24 hours postoperative
  Visual analogue score

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Hussien, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No